CLINICAL TRIAL: NCT00325676
Title: CONFIRM - Confirmation of Superiority of Complete Remission Concept Versus Classical Healing Concept for Treatment of Patients With Erosive GERD
Brief Title: Comparison of the Classical Healing Concept With the Complete Remission Concept After Treatment With Pantoprazole in Adult Patients With Erosive GERD (Gastroesophageal Reflux Disease) (BY1023/M3-342)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BY1023/M3-342
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2007-06

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; Pantoprazole; Complete Remission
MeSH Terms: conditions — Gastroesophageal Reflux; Pathologic Complete Response | interventions — Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole

SUMMARY:
The aim of this study is to evaluate the complete remission rates, endoscopic relapses, study discontinuation rates, and quality of life parameters in patients with erosive GERD. The study duration consists of a treatment period up to 16 weeks according to the classical healing concept or the complete remission concept. During this period, the patients will receive pantoprazole (tablet) at one dose level once daily. The following observational phase lasts up to 6 months. The study will provide further data on efficacy, safety, and tolerability of pantoprazole.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Endoscopically confirmed GERD (Los Angeles classification A-D)
* Patients whose compliance is expected to be high with respect to the completion of the questionnaires

Main Exclusion Criteria:

* Other gastrointestinal diseases
* Severe concomitant diseases
* Proton pump inhibitors (PPIs) during last 14 days before start
* H2 receptor antagonists, prokinetics during last 7 days before study start
* Helicobacter pylori (H. pylori) eradication during last 28 days before study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2006-06

PRIMARY OUTCOMES:
time to endoscopic relapse and/or unwillingness to continue due to GERD related symptoms

SECONDARY OUTCOMES:
further efficacy criteria
safety

CONTACTS AND LOCATIONS:
Overall Officials: Werner Janssen, MD, Principal Investigator — 23569 Lübeck, Germany
Locations (43):
- Brazil (13):
  - Altana Pharma/Nycomed, Belo Horizonte-MG
  - Altana Pharma/Nycomed, Blumenau - SC
  - Altana Pharma/Nycomed, Botucatu - SP
  - Altana Pharma/Nycomed, Campinas - Sao Paulo
  - Altana Pharma/Nycomed, Campinas - SP
  - Altana Pharma/Nycomed, Curitiba - PR
  - Altana Pharma/Nycomed, Ilha Do Fundao - Rio de Janeiro - RJ
  - Altana Pharma/Nycomed, Pinheiros Sao Paulo - SP
  - Altana Pharma/Nycomed, Porto Alegre - RS
  - Altana Pharma/Nycomed, Porto Alegre-RS
  - Altana Pharma/Nycomed, Ribeirao Preto-SP
  - Altana Pharma/Nycomed, Salvador-BA
  - Altana Pharma/Nycomed, São Paulo
- Germany (11):
  - Altana Pharma/Nycomed, Bad Schwalbach
  - Altana Pharma/Nycomed, Burg
  - Altana Pharma/Nycomed, Gardelegen
  - Altana Pharma/Nycomed, Königstein
  - Altana Pharma/Nycomed, Lübeck
  - Altana Pharma/Nycomed, Lüdenscheid
  - Altana Pharma/Nycomed, Lütjenburg
  - Altana Pharma/Nycomed, Nieder-Olm
  - Altana Pharma/Nycomed, Oelde
  - Altana Pharma/Nycomed, Wiesbaden
  - Altana Pharma/Nycomed, Wolmirstedt
- Poland (6):
  - Altana Pharma/Nycomed, Bydgoszcz
  - Altana Pharma/Nycomed, Inowrocław
  - Altana Pharma/Nycomed, Poznan
  - Altana Pharma/Nycomed, Siemianowice Śląskie
  - Altana Pharma/Nycomed, Torun
  - Altana Pharma/Nycomed, Tychy
- South Africa (13):
  - Altana Pharma/Nycomed, Berea, Durban
  - Altana Pharma/Nycomed, Bloemfontein
  - Altana Pharma/Nycomed, Cape Town
  - Altana Pharma/Nycomed, Durban
  - Altana Pharma/Nycomed, eManzimtoti
  - Altana Pharma/Nycomed, Goodwood
  - Altana Pharma/Nycomed, Johannesburg
  - Altana Pharma/Nycomed, Overport, Durban
  - Altana Pharma/Nycomed, Panorama
  - Altana Pharma/Nycomed, Pinetown
  - Altana Pharma/Nycomed, Port Elizabeth
  - Altana Pharma/Nycomed, Pretoria
  - Altana Pharma/Nycomed, Somerset West

REFERENCES:
- [Derived] Monnikes H, Schwan T, van Rensburg C, Straszak A, Theek C, Luhmann R, Sander P, Tholen A. Possible etiology of improvements in both quality of life and overlapping gastroesophageal reflux disease by proton pump inhibitor treatment in a prospective randomized controlled trial. BMC Gastroenterol. 2013 Oct 1;13:145. doi: 10.1186/1471-230X-13-145. PMID 24083350